CLINICAL TRIAL: NCT04001283
Title: Effect of Nitrite on Cardiac Muscle and Blood Vessels in Patients Undergoing Coronary Artery Bypass Grafting Surgery
Brief Title: Nitrite Effects on Cardiac Muscle in CABG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 87012
Record Dates: First submitted 2017-07-25; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Vascular Diseases; Cardiac Disease; Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Vascular Diseases; Heart Diseases; Diabetes Mellitus | interventions — Sodium Nitrite; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sodium nitrite 24hours before (Experimental): 10umol/min intravenous sodium nitrite for 30minutes at 1ml/min over a period of 30minutes, 24 hours prior to CABG surgery
  Interventions: Drug: Sodium Nitrite
- sodium nitrite 30minutes before (Experimental): 10umol/min intravenous sodium nitrite for 30minutes at 1ml/min over a period of 30minutes, 30 minutes prior to CABG surgery
  Interventions: Drug: Sodium Nitrite
- 0.9% sodium chloride (Placebo Comparator): Intravenous normal (0.9%) sodium chloride infused at 1ml/min
  Interventions: Drug: 0.9% Sodium-chloride

INTERVENTIONS:
Drug: Sodium Nitrite — Intravenous drug infusion
  Arms: sodium nitrite 24hours before; sodium nitrite 30minutes before
Drug: 0.9% Sodium-chloride — Matched placebo
  Arms: 0.9% sodium chloride

SUMMARY:
The purpose of this study is to test whether sodium nitrite affects the expression of cellular proteins important for metabolic and vascular function in vascular offcuts and cardiac biopsies taken from patients undergoing coronary artery bypass grafting (CABG) surgery.

DETAILED DESCRIPTION:
Nitrite has been shown in recent studies to improve cardiac performance, particularly in patients with heart failure. These improvements were demonstrated in measures that are independent of cardiac loading conditions, implying improved contractility via effects at a cellular level. In humans, coronary artery bypass graft (CABG) surgery presents an opportunity to safely obtain cardiac muscle biopsies and vascular tissue in order to investigate changes at a cellular level in these tissues.

The aim of this study is to investigate whether sodium nitrite affects the expression of cellular proteins important for heart muscle metabolism and vascular function when infused prior to routine CABG surgery. Patients undergoing CABG surgery who provide written informed consent will receive intravenous sodium nitrite 24hours prior to surgery, 30 minutes prior to surgery, or placebo. As Type 2 Diabetes Mellitus is common in patients undergoing CABG surgery, and itself has profound effects on metabolism, these patients will be sub-grouped into a diabetic cohort for interpretation of the molecular biology results. The 24hours prior to surgery vs. placebo arm will take place first, followed by the 30minutes prior to surgery vs. placebo arm. The data from this study will provide important information on the effects of nitrite on heart muscle and blood vessel tissues, and inform larger clinical trials in patients with cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

Males or females aged >18years scheduled to undergo coronary artery bypass grafting.

Exclusion Criteria:

Inability to read and understand the consent form and patient information leaflet Pregnancy and any woman of child bearing potential Patients with Type I diabetes Significant medical, surgical or psychiatric disease that in the opinion of the patient's attending physician would affect subject safety and participation in the trial including severe heart failure (NYHAIII-IV and EF<40%) and severe renal impairment (requiring dialysis).

Unstable coronary syndrome (within 2 weeks) Known glucose-6-phosphate dehydrogenase (G6PD) deficiency or G6PD deficiency measured at screening in males of African, Asian or Mediterranean decent.

Receipt of an investigational drug or biological agent within the 4 weeks prior to study entry or 5 times the drug half-life, whichever is the longer.

Intended heart valve surgery or additional surgery or redo-CABG surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2013-01-21 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic protein expression in cardiac biopsies and vascular offcuts | Taken during CABG surgery
  Cellular proteins that are important for metabolic regulation and vascular function that may be affected by nitrite such as eNOS, AKT, PDH

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Frenneaux, MD, FRCP, Principal Investigator — Clinical Professor, Norwich Medical School, The University of East Anglia, UK
Locations (2):
- United Kingdom (2):
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Papworth Hospital, Cambridge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ntessalen M, Procter NEK, Schwarz K, Loudon BL, Minnion M, Fernandez BO, Vassiliou VS, Vauzour D, Madhani M, Constantin-Teodosiu D, Horowitz JD, Feelisch M, Dawson D, Crichton PG, Frenneaux MP. Inorganic nitrate and nitrite supplementation fails to improve skeletal muscle mitochondrial efficiency in mice and humans. Am J Clin Nutr. 2020 Jan 1;111(1):79-89. doi: 10.1093/ajcn/nqz245. PMID 31599928